CLINICAL TRIAL: NCT01389089
Title: Effective Treatment of Posttraumatic and Postoperative Edema in Patients With Ankle- and Hindfoot Fractures. A Randomized Controlled Trial Comparing Multi-layer Compression Therapy and A-V Impulse Compression to the Standard Treatment With Ice
Brief Title: Effective Treatment of Posttraumatic and Postoperative Edema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Luzerner Kantonsspital (Other)
Collaborators: Orthofix Inc. (Industry); Medtronic - MITG (Industry)
Responsible Party: Principal Investigator, Reto Babst, Prof. Dr. med. Reto Babst, Senior Consultant Orthopedic Trauma, Luzerner Kantonsspital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 616
Record Dates: First submitted 2011-06-23; First posted 2011-07-07 (Estimated); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Edema
Keywords: edema reduction; ice; multi-layer compression bandage; A-V Impulse compression; ankle
MeSH Terms: conditions — Edema

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control group (Sham Comparator): The Control group received ice gel packs and elevation to reduce edema.
  Interventions: Behavioral: ice gel pack
- Multi-layer compression bandage (Experimental): A multi-layer compression bandage was applied to the lower limb and foot of the patient to reduce edema. Additionally, the limb was constantly elevated.
  Interventions: Other: Multi-layer compression bandage
- A-V Impulse compression (Active Comparator): An A-V Impulse compression device was used to reduce edema.
  Interventions: Device: A-V Impulse compression

INTERVENTIONS:
Behavioral: ice gel pack — ice gel pack combined with elevation
  Arms: Control group
Other: Multi-layer compression bandage — Application of a multi-layer compression bandage to the foot and lower limb (two layers of wool followed by several layers of a short stretch bandage).
  Other Names: Artiflex; Comprilan
  Arms: Multi-layer compression bandage
Device: A-V Impulse compression — A-V Impulse compression dosage: 130mmHg exerted to the sole of the foot for one second, every twenty second.
  Other Names: A-V intermittent Impulse compression device.; AVI
  Arms: A-V Impulse compression

SUMMARY:
Edema control after ankle- and hindfoot fractures is important. Multi-layer compression bandages or A-V Impulse compression may are more effective in reducing edema than ice.

DETAILED DESCRIPTION:
After ankle- and hindfoot fractures, edema has a major impact on the time point of surgical intervention and may increases the risk of wound complications and infection postoperatively. Effective treatment of edema, therefore, is of great importance. The aim of this study was to evaluate the efficacy of the multi-layer compression therapy and of the A-V Impulse compression (AVI) in reducing ankle- and hindfoot edema as compared to the standard treatment with ice.

ELIGIBILITY:
Inclusion criteria:

* Age 18-65 years
* Inpatients
* Acute ankle- or hindfoot fractures (malleolar-, calcaneus-, talus-, and pilon- tibial fractures) including fractures temporary stabilized with an external fixator)
* No walking aids before trauma
* Written informed consent
* Monotrauma
* Preoperative and/or postoperative edema
* Preoperative inclusion

  * if delay of surgery due to ankle edema
  * if fracture stable enough for temporary removal of orthesis

Exclusion criteria:

* Diabetes Mellitus
* Lymphedema
* Peripheral arterial occlusive disease (PAD)
* Decompensated heart failure or renal insufficiency
* Acute bacterial infection
* Severe osteoporosis
* Pathological fractures
* Known tumors
* Postthrombotic syndrome
* Thrombosis
* Open fractures
* Polytrauma, cerebral trauma
* Neurological deficiencies
* Diuretics
* Pregnancy
* Alcohol or drug abuse
* Psychological disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2007-01; Primary Completion 2009-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Ankle edema as measured with the figure-of-eight20 method | Participants were assessed daily for the duration of hospital stay, an expected average of 5 days preoperative and 5 days postoperative. Follow-up at 6 weeks postoperative.
  The figure-of-eight20 is a validated method to measure ankle edema with a simple spring tape. The spring tape follows a figure of eight around the ankle joint.

SECONDARY OUTCOMES:
Pain scores measured on the Visual Analogue Scale (VAS) | Participants were assessed daily for the duration of hospital stay, an expected average of 5 days preoperative and 5 days postoperative. Follow-ups at 6 weeks, 12 weeks and 1 year postoperative.
  Visual Analogue Scales were used to assess a daily pain score reflecting strongest and average pain perceived during the previous 24 hours, night pain and pain frequency.
Patient satisfaction with treatment scores measured on the Visual Analogue Scale | Participants were assessed for the duration of hospital stay, an expected average of 5 days preoperative and 5 days postoperative --> assessment at the day of discharge.
  Visual Analogue Scales were used to assess patient satisfaction with the assigned treatment. The patients had to record their satisfaction with the treatment before surgery and after surgery.
Number of days until possible operation | Participants were assessed daily for the duration of preoperative hospital stay, an expected average of 5 days.
  The surgeon daily had to assess whether the patient was ready for operation or not. The wrinkling test served as a criteria for decision making. Accordingly the number of days until possible operation was recorded.
Number of postoperative hospitalization days | Participants were assessed daily for the duration of postoperative hospital stay, an expected average of 5 days.
  Postoperatively the physiotherapist each day had to record whether or not the patient was ready for discharge. Discharge criteria: 1. patient is able to walk 20 meters and one flight of stairs with crutches. 2. the wound is dry and not irritated. Accordingly, the number of days of postoperative hospitalization until discharge criteria were reached was recorded.
Range of motion of the ankle joint and foot. | Participants were assessed daily for the duration of postoperative hospital stay, an expected average of 5 days. Follow-up at 6 weeks postoperative.
  Plantar flexion, dorsal flexion, inversion and eversion were assessed with a hydrogoniometer.
Amount of daily intake of medication | Participants were assessed daily for the duration of hospital stay, an expected average of 5 days preoperative and 5 days postoperative.
  The intake of daily pain medication was recorded for the instay period (Dafalgan, Novalgin, opiates). Furthermore, the patient file was screened for any Nonsteroidal anti-inflammatory drugs (not allowed).
Number of adverse events as a measure of safety in each group | Participants were assessed daily for the duration of hospital stay, an expected average of 5 days preoperative and 5 days postoperative. Patient file was screened for adverse events until 1 year postoperatively.
  Adverse events were defined as:
  bacterial infection, implant breakage, secondary dislocations, massive wound complications, thrombosis, embolism.
Lower limb function (Foot and ankle ability measure) | 12 weeks postoperative, 1 year postoperative.
  Questionnaire, self-assessed by the patient. To assess function and participation.
General Health (SF-36) | 12 weeks postoperative,1 year postoperative.
  Generic assessment of the health status with the SF-36.
Patient satisfaction scores on overall outcome measured on the Visual Analogue Scale | 12 weeks and 1 year postoperative.
  Patients had to record on the VAS on how satisfied they were with the overall outcome.
Amount of volumetric lower limb edema | Participants were assessed daily for the duration of hospital stay, an expected average of 5 days preoperative and 5 days postoperative. Follow-up at 6 weeks postoperative.
  Measurements of circumference of the lower limb were used to calculate lower limb volume. The circumferences of the lower limb were measured in increments of 4 cm from ankle level until below the knee joint.
Number of complains of discomfort or intolerances considering the intervention | Participants were assessed daily for the duration of hospital stay, an expected average of 5 days preoperative and 5 days postoperative.
  Every day the patients were asked by the physiotherapist if they had any sort of complains considering the assigned treatment (discomfort or intolerances).

CONTACTS AND LOCATIONS:
Overall Officials: Reto Babst, Prof.Dr.med., Principal Investigator — Luzerner Kantonsspital
Locations (1):
- Luzerner Kantonsspital, Unfallchirurgie, Lucerne, Switzerland